CLINICAL TRIAL: NCT02507440
Title: Impact of Topical Pharyngeal Anesthetics on Discharge of the Patients When Used in Conjunction With Propofol Sedation in Routine EGD's
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bassett Healthcare (Other)
Responsible Party: Principal Investigator, David A Ullman MD, Attending Physician - Anesthesiology, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Topical Anesthesia
MeSH Terms: interventions — Lidocaine; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viscous Lidocaine (Active Comparator): Five minutes prior to intravenous sedation the patients will be asked to gargle with 7.5 ml of 2% lidocaine viscous solution and swallow.
  Interventions: Drug: Lidocaine; Drug: Propofol
- Placebo (Placebo Comparator): Five minutes prior to intravenous sedation the patients will be asked to gargle with 7.5 ml of placebo and then swallow. Placebo will be 3% methylcellulose which will be flavored and colored to match the characteristics of 2 % lidocaine.
  Interventions: Drug: Placebo; Drug: Propofol

INTERVENTIONS:
Drug: Lidocaine — Prior to initiation of anesthesia viscous lidocaine or placebo will be administered.
  Arms: Viscous Lidocaine
Drug: Placebo — Prior to initiation of anesthesia viscous lidocaine or placebo will be administered.
  Arms: Placebo
Drug: Propofol — All patients will receive intravenous propofol as anesthesia for EGD

SUMMARY:
To find out if the administration of the local pharyngeal anesthetic, lidocaine, in conjunction with Propofol during elective Esophagogastroduodenoscopy (EGD) is useful, safe and impacts the time of discharge of patient compared to placebo.

DETAILED DESCRIPTION:
Local pharyngeal anesthetics when used in conjunction with IV sedatives such as benzodiazepines may ease the endoscopy and the patient tolerance. They have been believed to dull the gag reflex and smooth the process of intubation of the esophagus. However local pharyngeal anesthetics beside increasing the total procedure time and delaying the discharge of the patient can cause serious side effects including methemoglobinemia, aspiration and anaphylactic reactions although these are rare. There have been studies supporting the use of local pharyngeal anesthetics along with sedatives such as benzodiazepines and opiates [1]. However there have been only a few studies on the use of local pharyngeal anesthetics in conjunction with propofol which have not supported any added benefit of local pharyngeal anesthetics [2, 3, 4]. Despite of these studies local pharyngeal anesthetics are still being widely used in conjunction with propofol during EGD's. There are currently no set recommendations or protocol for the use of local anesthetics such as lidocaine in conjunction with propofol during EGD's. This study is yet another attempt to find out if the local pharyngeal anesthetics have any role during EGD's when used in conjunction with propofol.

This will be a randomized, double blind, placebo controlled trial. Patients scheduled to have elective EGD's will be consented for their participation. CRNA's or anesthetists would be present during all EGD's since propofol is only given by the anesthesia department personnel. Five minutes prior to intravenous sedation the patients will be asked to gargle with 7.5 ml of 2% lidocaine viscous solution or 7.5 ml of placebo and then swallow. Placebo will be 3% methylcellulose which will be flavored and colored to match the characteristics of 2 % lidocaine. The operating gastroenterologist after extubation will be asked to fill in a questionnaire commenting on the ease of intubation and if they were able to make any guesses whether lidocaine was used during the procedure or not. An independent observer will be asked to fill in a questionnaire regarding their visual assessment about patient discomfort during the procedure. the visual scale ranging from 1 cm to 10 cm and then the observer; gastroenterologist would pick up a number with 0 being the worst satisfaction and 10 being the best satisfaction with the procedure. The questionnaire will also include the number of times the patient gagged, number of intubation attempts by the gastroenterologist and post procedure what did the gastroenterologist think if Lidocaine or placebo was used during the procedure. The time after recovery from the sedatives till the patient is discharged will be recorded as the primary end point. The total number of intubation attempts, total amount of propofol used during the procedure and any above mentioned side effects of lidocaine will be recorded as the secondary end points. The total procedure time will also be recorded. Start time for the procedure will be when the first attempt for GI scope insertion is made by the gastroenterologist after giving sedative. End time for the procedure is when the GI scope is extubated. Throat pain/discomfort scores which are routinely assessed and recorded prior to discharge will be assessed as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older.
* Scheduled for an elective EGD.

Exclusion Criteria:

* Patients having EGD for urgent or emergent reasons.
* Patients having therapeutic EGD's.
* History of intolerance to either lidocaine or propofol.
* Pregnancy.
* Impaired swallowing reflex.
* Dementia
* Patients unable to consent on own for the procedure and/or research.
* Patient receiving any other sedative in addition to Propofol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Time from study drug administration to discharge | 3 hours
  The time from study drug administration to discharge from procedure area will be measured.

SECONDARY OUTCOMES:
Gastroenterologist satisfaction at time of intubation | 15 minutes
  Gastroenterologist performing the EGD will complete a 10 cm VAS scale indicating satisfaction with ease of intubation.
Propofol dose | 30 minutes
  total propofol dose administered during the procedure will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: david Ullman, MD, Principal Investigator — Bassett Healthcare
Locations (1):
- Bassett Healthcare Network, Cooperstown, New York, United States